CLINICAL TRIAL: NCT03295201
Title: Clinical Effects of Exercise Program Added to Pulmonary Rehabilitation in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09.2015.287
Record Dates: First submitted 2017-08-23; First posted 2017-09-27 (Actual); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Postural exercise; Pulmonary rehabilitation
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary rehabilitation+exercise group (Experimental): Active cycle of breathing techniques (ACBT) and postural exercise program
  Interventions: Other: Active cycle of breathing techniques (ACBT); Other: Postural Exercise
- Pulmonary rehabilitation group (Active Comparator): Active cycle of breathing techniques (ACBT)
  Interventions: Other: Active cycle of breathing techniques (ACBT)

INTERVENTIONS:
Other: Active cycle of breathing techniques (ACBT) — ACBT involves three phases (Breathing control, chest expansion exercise, and huff coughing). These phases will apply with a sequence to remove secretion. ACBT will apply 1 per a week for 6 weeks.
Other: Postural Exercise — Postural exercise program will include thoracic vertebra mobilization, pectoral stretching, scapula and thoracic extensors strengthening and core stability exercises. Postural exercise program will apply 1 per a week for 6 weeks.
  Arms: Pulmonary rehabilitation+exercise group

SUMMARY:
The aim of this study is to investigate the effects of postural exercise program added to pulmonary rehabilitation program on quality of life, exercise tolerance and postural stability in children with Cystic Fibrosis.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an autosomal recessive, multisystem involvement disease. The most important cause of mortality in CF is pulmonary complications. Prevention of pulmonary complications is only possible with pulmonary rehabilitation. Pulmonary rehabilitation methods used in CF are called airway cleaning techniques that include postural drainage, breathing techniques and use of devices. These techniques have not been proven to be superior to each other. Active cycle of breathing techniques (ACBT) is one of the breathing techniques used to remove secretions from the lungs.

Pulmonary disease progression in CF causes postural impairment and decrease of exercise tolerance, which can reduce effectiveness of pulmonary rehabilitation. The aim of this study is to investigate the effects of postural exercise program added to pulmonary rehabilitation program on quality of life, exercise tolerance and postural stability in children with CF.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed with KF
2. Be able to understand commands

Exclusion Criteria:

1. FEV1 below than %30
2. Cor pulmonale
3. Advanced gastroesophageal reflux
4. Current hospital admission due to lung infection
5. Be diagnosed with neuromuscular disease

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag Saygi, MD, Prof, Study Director — Marmara University School of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Marmara University School of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edwards J, Clarke A, Greenop D. Adults with cystic fibrosis - responding to a new ageing population. Chronic Illn. 2013 Dec;9(4):312-9. doi: 10.1177/1742395313479982. Epub 2013 May 23. PMID 23702786
- [Background] Barker N, Raghavan A, Buttling P, Douros K, Everard ML. Thoracic Kyphosis is Now Uncommon Amongst Children and Adolescents with Cystic Fibrosis. Front Pediatr. 2014 Feb 17;2:11. doi: 10.3389/fped.2014.00011. eCollection 2014. PMID 24596827
- [Background] Tattersall R, Walshaw MJ. Posture and cystic fibrosis. J R Soc Med. 2003;96 Suppl 43(Suppl 43):18-22. No abstract available. PMID 12906321
- [Background] Daniels T. Physiotherapeutic management strategies for the treatment of cystic fibrosis in adults. J Multidiscip Healthc. 2010 Nov 19;3:201-12. doi: 10.2147/JMDH.S8878. PMID 21289861
- [Background] Massery M. Musculoskeletal and neuromuscular interventions: a physical approach to cystic fibrosis. J R Soc Med. 2005;98 Suppl 45(Suppl 45):55-66. PMID 16025768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was March 2017-October 2017 Setting: A university hospital outpatient clinics
Pre-assignment Details: Number of patients assessed for eligibility was 30. Among them,8 participants were excluded due to being inappropiate for the inclusion criteria (6 were out of age limits, 2 did not agree to participate in the study)
Period: Overall Study
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Started | 11 | 11
Completed | 10 | 9
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Hospital admission | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (2) | 10 (3) | 9 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 10 | 9 | 19
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 16 (2) | 16 (2) | 16 (2)

OUTCOME MEASURES:

1. Primary Outcome: Exercise Tolerance
Description: Modified Shuttle Test (MST) is used to measure the exercise tolerance. The patient is asked to walk until feeling tired between two fixed objects with a 10-meter interval, starting at normal walking speed and increasing the speed at the beginning of each minute. Maximum distance (meters) is measured for the test.
Time Frame: Before treatment
Measure: Mean (Standard Error); unit: meters
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
meters | 817 (234.62) | 792.22 (327.21)

2. Primary Outcome: Exercise Tolerance
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: meters
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
meters | 980 (277.24) | 1058.77 (594.67)

3. Primary Outcome: Exercise Tolerance
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Error); unit: meters
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
meters | 1104 (306.73) | 1036.66 (457.16)

4. Primary Outcome: Exercise Tolerance
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Error); unit: meters
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
meters | 1251 (324.15) | 1161.11 (594.06)

5. Secondary Outcome: Quality of Life
Description: The Cystic Fibrosis Questionnaire-Revised (CFQR) is used to measure the quality of life. This scale is found to be valid and reliable in Turkish. The child version of this test consists 35 questions about physical function, emotional function, social function, body appearance, eating disorders, treatment difficulties, respiratory and digestive symptoms. The total score is calculated between 0-100 and higher scores define the better condition.
Time Frame: Before treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
units on a scale | 86.4 (5.75) | 92.77 (9.94)

6. Secondary Outcome: Quality of Life
Description: as for outcome 5
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
units on a scale | 88.9 (7.04) | 90.88 (13.37)

7. Secondary Outcome: Quality of Life
Description: as for outcome 5
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
units on a scale | 87.2 (5.57) | 93.33 (11.35)

8. Secondary Outcome: Quality of Life
Description: as for outcome 5
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
units on a scale | 89.7 (7.84) | 95.55 (12.64)

9. Secondary Outcome: Postural Stability
Description: The Balance Master Device- Limits of Stability Test (LOS) is used for to measure the postural stability of children. The LOS consists a 18x60 inch of a pressure platform which connected to a computer system. The patient is asked to stand on the platform barefoot and watch the image which can be moved by trunk movement on the computer the monitor. It is required to move the image towards to target points on the monitor with commands. Reaction time, movement velocity, endpoint excursion, maximum excursion and direction control parameters are calculated during these trunk movements. Reaction time (seconds) parameter is preferred to use for this study.
Time Frame: Before treatment
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
seconds | 1.29 (0.85) | 1.03 (0.53)

10. Secondary Outcome: Postural Stability
Description: as for outcome 9
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
seconds | 0.91 (0.66) | 0.83 (0.65)

11. Secondary Outcome: Postural Stability
Description: as for outcome 9
Time Frame: 3 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
seconds | 0.88 (0.72) | 0.65 (0.52)

12. Secondary Outcome: Postural Stability
Description: as for outcome 9
Time Frame: 6 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
seconds | 1.15 (0.69) | 0.92 (0.46)

13. Secondary Outcome: Pulmonary Function
Description: Forced expiratory volume in 1 second (FEV1)
Time Frame: Before treatment
Measure: Mean (Standard Deviation); unit: millilitres
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
millilitres | 82.8 (14.57) | 83.78 (21.06)

14. Secondary Outcome: Pulmonary Function
Description: Forced expiratory volume in 1 second (FEV1)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: millilitres
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
millilitres | 93.3 (21.71) | 82.11 (17.14)

15. Secondary Outcome: Pulmonary Function
Description: Forced expiratory volume in 1 second (FEV1)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: millilitres
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
millilitres | 86.6 (12.19) | 82.77 (17.85)

16. Secondary Outcome: Pulmonary Function
Description: Forced expiratory volume in 1 second (FEV1)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: millilitres
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
millilitres | 87.7 (16.95) | 90 (23.52)

17. Secondary Outcome: Spinal Deformity- The Cobb Angle (Researcher 1)
Description: The Cobb angle was measured on anteroposterior scoliosis graphs by the angle between the superior end plate of the vertebra corpus where the curve begins and the end plate of the vertebra corpus which the curve ends.
Time Frame: Before treatment
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
degrees | 2.37 (1.40) | 7.75 (5.95)

18. Secondary Outcome: Spinal Deformity- The Cobb Angle (Researcher 2)
Description: as for outcome 17
Time Frame: Before treatment
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
degrees | 2.12 (2.1) | 7.75 (5.12)

19. Secondary Outcome: Spinal Deformity- The Cobb Angle (Researcher 1)
Description: as for outcome 17
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
degrees | 3.5 (2.56) | 5.25 (3.41)

20. Secondary Outcome: Spinal Deformity- The Cobb Angle (Researcher 2)
Description: as for outcome 17
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
degrees | 3.88 (2.42) | 5.5 (2.83)

21. Secondary Outcome: Spinal Deformity- The Modified Cobb Angle (Researcher 1)
Description: The Modified Cobb angle was found on lateral scoliosis graphs by the angle between the superior end plate of the T4 vertebra corpus and the inferior end plate of the T12 vertebra corpus.
Time Frame: Before treatment
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
degrees | 35.33 (12.62) | 34.33 (6.84)

22. Secondary Outcome: Spinal Deformity- The Modified Cobb Angle (Researcher 2)
Description: as for outcome 21
Time Frame: Before treatment
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
degrees | 34.67 (11.76) | 33.11 (7.4)

23. Secondary Outcome: Spinal Deformity- The Modified Cobb Angle (Researcher 1)
Description: as for outcome 21
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
degrees | 35.5 (8.09) | 32.33 (3.08)

24. Secondary Outcome: Spinal Deformity- The Modified Cobb Angle (Researcher 2)
Description: as for outcome 21
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
Number analyzed (Participants) | 10 | 9
degrees | 35 (7.87) | 32.4 (3.33)

ADVERSE EVENTS:
Time Frame: 6 months
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored.
Arm/Group | Pulmonary Rehabilitation+Exercise Group | Pulmonary Rehabilitation Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT03295201/Prot_SAP_000.pdf